CLINICAL TRIAL: NCT07287150
Title: A Phase II, Randomized, Multicenter, Open-Label Study Evaluating the Efficacy and Safety of the Combination of Inavolisib Plus Enzalutamide Versus Physician's Choice of ARPI or Docetaxel in Patients With Metastatis Castration-Resistant Prostate Cancer
Brief Title: A Study to Test Inavolisib Treatment in Participants With Metastatic Castration-Resistant Prostate Cancer
Acronym: InavoPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO45813; 2025-521327-67-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-11; First posted 2025-12-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
MeSH Terms: interventions — inavolisib; enzalutamide; abiraterone; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm 1 (Experimental): Participants will receive Inavolisib plus enzalutamide
  Interventions: Drug: Inavolisib; Drug: Enzalutamide; Diagnostic Test: FoundationOne® CDx (F1CDx) Assay
- Arm 2 (Active Comparator): Participants will receive either ARPi switch (enzalutamide or abiraterone) or docetaxel
  Interventions: Drug: Enzalutamide; Drug: Abiraterone; Drug: Docetaxel; Diagnostic Test: FoundationOne® CDx (F1CDx) Assay

INTERVENTIONS:
Drug: Inavolisib — Inavolisib will be administered orally as per the schedule specified in the protocol.
  Arms: Arm 1
Drug: Enzalutamide — Enzalutamide will be administered orally as per the schedule specified in the protocol.
Drug: Abiraterone — Abiraterone will be administered orally as per the schedule specified in the protocol.
  Arms: Arm 2
Drug: Docetaxel — Docetaxel will be administered intravenously as per the schedule specified in the protocol.
  Arms: Arm 2
Diagnostic Test: FoundationOne® CDx (F1CDx) Assay — F1CDx is a next-generation sequencing (NGS)-based in vitro diagnostic test that will be used to determine a participant's biomarker status.

SUMMARY:
This study will evaluate the efficacy and safety of the combination of inavolisib plus enzalutamide compared with physician's choice of alternative androgen receptor pathway inhibitor (ARPi) or docetaxel in biomarker-selected participants with metastatic castrate-resistant prostate cancer (mCRPC) who have received one prior second-generation ARPi.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without small-cell or neuroendocrine features
* Progressive metastatic CRPC, defined as any of the following: PSA progression, defined by a minimum of two rising PSA values from three consecutive assessments with an interval of at least 7 days between assessments and with a minimal starting value of PSA >=1 ng/mL; The most recent qualifying PSA value must be determined within 14 days of enrollment; Soft tissue disease progression, defined by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1); Bone disease progression, defined by PCWG3 criteria, with two or more new metastatic bone lesions on a whole-body radionuclide bone scan
* Treatment with at least one, but no more than one, prior second-generation ARPi (abiraterone, apalutamide, enzalutamide, darolutamide) for hormone- sensitive prostate cancer (HSPC) or CRPC
* Availability of a tumor tissue specimen that is suitable (e.g., adequate quality and quantity) for use in determining biomarker status
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Fasting glucose </= 100 mg/dL and HbA1c < 5.7%

Exclusion Criteria:

* Presence of liver metastasis
* Prior treatment with any phosphatidylinositol-3-kinase (PI3K), protein kinase B (AKT), or mammalian target of rapamycin (mTOR) inhibitor, or with any agent with a mechanism of action of inhibiting the PI3K/AKT/mTOR pathway
* Type 1 or Type 2 diabetes mellitus
* Prior treatment for mCRPC with cytotoxic chemotherapy or novel hormonal treatments (e.g., androgen receptor degraders, CYP11 inhibitors), with the following treatments permitted: Prior docetaxel in mHSPC, providing no evidence of disease progression occurred during treatment or within 6 months of treatment completion; Prior docetaxel in the adjuvant or neoadjuvant setting providing no evidence of disease progression occurred during treatment or within 12 months of treatment completion; Prior treatment with sipuleucel-T, with the last dose administered >28 days prior to start of treatment; Prior PARPi therapy, as per local prescribing information, with the last dose administered >14 days prior to start of treatment; One prior RLT or radiotherapeutic agent (e.g., PSMA-targeted RLT, Radium 223) with the last dose administered >8 weeks prior to start of treatment
* One prior RLT or radiotherapeutic agent (e.g., PSMA-targeted RLT, Radium 223) with the last dose administered > 8 weeks prior to start of treatment
* Other concurrent anti-cancer therapy except for androgen deprivation therapy
* Treatment with strong CYP2C8 inhibitors, strong or moderate CYP2C8 inducers, or strong CYP3A4 inducers within 1 week or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study treatment
* Transfusion of any blood product for the sole purpose of making a potential participant eligible for study inclusion or within 28 days of enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-05-14 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-free Survival (rPFS) | Up to approximately 5 years

SECONDARY OUTCOMES:
Percentage of Participants with Confirmed Composite Response Rate (RR) | Up to approximately 5 years
Percentage of Participants with Confirmed Prostate-Specific Antigen 90 (PSA90) | Up to approximately 5 years
Percentage of Participants with Confirmed Prostate-Specific Antigen 50 (PSA50) | Up to approximately 5 years
Objective Response Rate (ORR) | Up to approximately 5 years
Duration of Response (DOR) | Up to approximately 5 years
Overall Survival (OS) | Up to approximately 5 years
Percentage of Participants With Adverse Events (AEs) | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (2):
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- Jewish General Hospital, Montreal, Quebec, Canada
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing